CLINICAL TRIAL: NCT00492115
Title: Cognitive Benefits of Treating Sleep Apnea in Dementia
Brief Title: Cognitive Benefits of Treating Sleep Apnea in Parkinson's Disease
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sonia Ancoli-Israel, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG08415; R01AG008415 (NIH)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Parkinson's Disease; Sleep Disordered Breathing
Keywords: sleep; dementia; apnea; memory; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Sleep Apnea Syndromes; Dementia; Apnea | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- therapeutic CPAP Treatment (6 weeks)" (Active Comparator): Intervention - The active comparator is an intervention of nightly therapeutic CPAP (continuous positive airway pressure) treatment for 6 weeks. Patients will use CPAP every night for the full duration of the study, i.e., 6 weeks
  Interventions: Device: Continuous positive airway pressure (CPAP)
- Sham CPAP/therapetuic CPAP (6 weeks)" (Placebo Comparator): The placebo comparator is an intervention of placebo CPAP (continuous positive airway pressure) nightly for 3 weeks followed by therapeutic CPAP treatment nightly for 3 weeks.
  Patients will use a sham CPAP (no real pressure) for 3 weeks and then will be switched to real CPAP for 3 weeks.
  Interventions: Device: Placebo CPAP

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — therapeutic Continuous positive airway pressure (tCPAP) nightly for 6 weeks
  Arms: therapeutic CPAP Treatment (6 weeks)"
Device: Placebo CPAP — Ineffective Continuous positive airway pressure (pCPAP) for 3 weeks followed by therapeutic CPAP for 3 weeks
  Arms: Sham CPAP/therapetuic CPAP (6 weeks)"

SUMMARY:
Patients with sleep disordered breathing (SDB), also called sleep apnea, experience nighttime disrupted sleep and, because they stop breathing for short periods during the night, do not get sufficient oxygen to their brains. This can frequently result in daytime impairments including difficulties with memory. The state-of-the-art treatment for SDB is Continuous Positive Airway Pressure (CPAP). Many non-demented SDB patients who are successfully treated with CPAP show improvement in memory and other cognitive functions. Data have shown that patients with Parkinson's disease have a high rate of SDB. Patients with Parkinson's disease also often have problems with memory. This study will test the effects of treating SDB among patients with Parkinson's disease and SDB. Specifically, the study will test the effect of CPAP treatment on SDB and sleep; the effect of CPAP treatment on daytime sleepiness, cognition, overall quality of life and mood; the effect of CPAP treatment on the frequency of symptoms of REM behavior disorder and restless legs syndrome; the effect of continued CPAP use (beyond the six weeks of the study) on SDB, sleep, cognition, mood and quality of life; whether the study-partner feels that CPAP improves the patient's sleep, mood and overall functioning; whether study-partners feel that their own sleep, mood and overall functioning improve as the patient's sleep improves both during the 6-week protocol and at follow-up for those opting to continue using CPAP.

DETAILED DESCRIPTION:
This study will examine the effect of three weeks vs. six weeks of CPAP treatment on cognitive functioning and sleep in patients with Parkinson's disease and sleep apnea. It is designed as a randomized, double blind, placebo-controlled trial of CPAP. As a comparison group, half the patients will first be randomly assigned to three weeks of shamCPAP, followed by three weeks of therapeutic CPAP treatment. Sleep, functional outcome and mood questionnaires and a repeatable neuropsychological test battery, chosen to be sensitive to the type of changes we expect to find in memory and cognitive function, will be administered before the start of treatment, after three weeks, and after six weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of dementia due to Parkinson's disease (according to the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (code 294.1)
* MMSE score between 18 and 26, inclusive; cognitive symptoms must occur at least one year after the diagnosis of PDD
* Apnea hypopnea index >10 (i.e., 10 apneas plus hypopneas per hour of sleep)
* Over the age of 50 years
* Stable health
* Fluent English speaking
* Patients will be allowed to continue dopaminergic medications, acetylcholinesterase inhibitors, psychotropic medications, memory enhancers, health food supplements, etc. as long as they have been stable on the same dose for at least two months prior to participation and agree to continue on this dose for the duration of the 6-week study.

Exclusion Criteria:

* Current treatment for sleep apnea (to avoid discontinuing already established treatment for sleep apnea and any carry over confounding effect of treatment on cognition).
* Central sleep apnea
* Use of medications known to influence sleep (i.e. sedative hypnotics, narcotics) if the dose cannot remain stable for the duration of the study.
* Bronchospastic and symptomatic chronic obstructive pulmonary disease as indicated by regular use of bronchodilators, steroids, history of carbon dioxide retention, waking hypoxemia (PaO2 <60 mmHg or SpO2 <92 % by pulse oximetry), or use of supplemental oxygen.
* Symptomatic coronary or cerebral vascular disease (history of myocardial infarction, angina, stroke, or transient ischemic attacks), history of life-threatening arrhythmias, cardiomyopathy, or current alcohol or drug abuse
* Current diagnosis of active seizure disorder; presence of any neurodegenerative disorder other than PDD or other causes of dementia
* Any behavioral or physical problem that would preclude completion of the primary evaluation or treatment with CPAP.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Ancoli-Israel, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cooke JR, Liu L, Natarajan L, He F, Marler M, Loredo JS, Corey-Bloom J, Palmer BW, Greenfield D, Ancoli-Israel S. The effect of sleep-disordered breathing on stages of sleep in patients with Alzheimer's disease. Behav Sleep Med. 2006;4(4):219-27. doi: 10.1207/s15402010bsm0404_2. PMID 17083302
- [Result] Chong MS, Ayalon L, Marler M, Loredo JS, Corey-Bloom J, Palmer BW, Liu L, Ancoli-Israel S. Continuous positive airway pressure reduces subjective daytime sleepiness in patients with mild to moderate Alzheimer's disease with sleep disordered breathing. J Am Geriatr Soc. 2006 May;54(5):777-81. doi: 10.1111/j.1532-5415.2006.00694.x. PMID 16696743
- [Result] Ayalon L, Ancoli-Israel S, Stepnowsky C, Marler M, Palmer BW, Liu L, Loredo JS, Corey-Bloom J, Greenfield D, Cooke J. Adherence to continuous positive airway pressure treatment in patients with Alzheimer's disease and obstructive sleep apnea. Am J Geriatr Psychiatry. 2006 Feb;14(2):176-80. doi: 10.1097/01.JGP.0000192484.12684.cd. PMID 16473983
- [Derived] Harmell AL, Neikrug AB, Palmer BW, Avanzino JA, Liu L, Maglione JE, Natarajan L, Corey-Bloom J, Loredo JS, Ancoli-Israel S. Obstructive Sleep Apnea and Cognition in Parkinson's disease. Sleep Med. 2016 May;21:28-34. doi: 10.1016/j.sleep.2016.01.001. Epub 2016 Feb 10. PMID 27448468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were referred to UCSD by community neurologists or volunteered after hearing a talk about the study at PD support group meetings.
Pre-assignment Details: 183 contacted; 144 screened/phone; 106 consented, 5 dropped/12 excluded; 89 screened for apnea with sleep study (2 dropped during night study), 44 had no sleep apnea. 5 declined treatment.
  19 participants randomized to each arm
Groups:
- A: Continuous Positive Airway Pressure (CPAP): Continuous positive airway pressure (CPAP)
  Continuous positive airway pressure (CPAP): therapeutic CPAP for six weeks
- B: Placebo Continuous Positive Airway Pressure: Placebo Continuous Positive airway pressure
  Placebo CPAP: Ineffective CPAP 3 weeks placebo CPAP followed by 3 weeks of therapeutic CPAP
Period: Overall Study
Arm/Group | A: Continuous Positive Airway Pressure (CPAP) | B: Placebo Continuous Positive Airway Pressure
Started | 19 | 19
Completed | 16 (3 dropped due to anxiety or not being able to tolerate CPAP) | 15 (4 dropped due to not being able to tolerate CPAP)
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- A: Continuous Positive Airway Pressure: Continuous Positive Airway Pressure (therapeutic CPAP) for 6 weeks
- B. Sham CPAP: Sham (placebo) CPAP for 3 weeks followed by therapeutic CPAP for 3 weeks.
- Total: Total of all reporting groups
Arm/Group | A: Continuous Positive Airway Pressure | B. Sham CPAP | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.5) | 67.7 (10.0) | 67.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Tests to Determine the Apnea-hypopnea Index (Number of Apneas and Hypopneas Per Hour of Sleep)
Description: Overnight sleep studies were done to determine the effect of treatment on the apnea-hypopnea index (number of apneas and hypopneas per hour of sleep)
Time Frame: six weeks
Measure: Mean (Standard Deviation); unit: apnea hypopnea index
Groups:
- A: Continuous Positive Airway Pressure (CPAP):: CPAP
  Continuous positive airway pressure (CPAP): therapeutic CPAP
- B: Placebo CPAP: Ineffective CPAP: Placebo CPAP
  Placebo CPAP: Ineffective CPAP
Arm/Group | A: Continuous Positive Airway Pressure (CPAP): | B: Placebo CPAP: Ineffective CPAP
Number analyzed (Participants) | 17 | 15
apnea hypopnea index | 5.2 (2) | 20 (4)

2. Secondary Outcome: Sleep Stages; %Time Spent at SaO2<90%;
Description: Overnight sleep studies were done to examine the effect of CPAP treatment on sleep stages and on %time spent at Sa)2<90%.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percent time spent at low oxygen <90%
Arm/Group | A: Continuous Positive Airway Pressure (CPAP): | B: Placebo CPAP: Ineffective CPAP
Number analyzed (Participants) | 17 | 15
Percent time spent at low oxygen <90% | 2.1 (1) | 12.9 (5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the full 6 weeks per participant
Groups:
- A: Continuous Positive Airway Pressure (CPAP): Therapeutic CPA: CPAP
  Continuous positive airway pressure (CPAP): therapeutic CPAP for 6 weeks
- B: Placebo CPAP: Ineffective CPAP: Placebo CPAP
  Placebo CPAP: Ineffective CPAP for 3 weeks followed by therapeutic CPAP for 3 weeks
Arm/Group | A: Continuous Positive Airway Pressure (CPAP): Therapeutic CPA | B: Placebo CPAP: Ineffective CPAP
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No